CLINICAL TRIAL: NCT05145764
Title: Suvorexant as an Adjunct to Buprenorphine Induction and Maintenance in Persons Who Use Fentanyl
Brief Title: Suvorexant as an Adjunct to Buprenorphine in Persons Who Use Fentanyl
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00301337; UH3DA048734 (NIH)
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Suvorexant; Placebo; Opioid Use Disorder
Keywords: Opioid use disorder; Insomnia; Suvorexant; Fentanyl; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suvorexant (Experimental): Nightly dosing of suvorexant
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): Nightly dosing of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — Encapsulated suvorexant (matched for color, weight, and size)
  Arms: Suvorexant
Drug: Placebo — Encapsulated placebo (matched for color, weight, and size)
  Arms: Placebo

SUMMARY:
This is a 4-week, randomized-controlled trial of suvorexant vs placebo in persons with opioid use disorder who have recent fentanyl exposure. Participants will first undergo a 5-day residential phase wherein participants are stabilized on sublingual buprenorphine/naloxone, followed by a 3-week outpatient phase wherein participants are maintained on sublingual buprenorphine/naloxone and transitioned to extended-release buprenorphine).

DETAILED DESCRIPTION:
This study will enroll persons with opioid use disorder (N=120) who have recent fentanyl exposure (as assessed via urinalysis testing). Participants will be randomized to receive suvorexant or placebo for the duration of the study enrollment, which will serve as the between-groups experimental comparison. The study will consist of a brief (5 day) residential phase and 3-week outpatient phase. During the residential phase, all participants will be briefly maintained on a short acting opioid prior to induction onto sublingual (SL) buprenorphine (using either the buprenorphine or buprenorphine/naloxone product). At the end of the 5-day residential period, participants will be discharged to complete the ~3-week outpatient phase. During the outpatient period all participants will be maintained on SL buprenorphine/naloxone and continue to receive suvorexant or placebo, and at the end of the study participants will receive an injection of XR-buprenorphine (Sublocade). All buprenorphine procedures will be open label and will follow standard-of-care practices. Study medication during the outpatient period will be managed using an automated pill dispenser. Data collection will consist of forehead-based EEG monitoring, wrist-worn actigraphy/photoplethysmography, and questionnaires delivered during study visits or via cell-phone based ecological momentary assessments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Meets DSM-5 criteria for opioid use disorder (OUD) with evidence of physical dependence on opioids
* Provides a urine sample that tests positive for fentanyl and/or fentanyl analogues
* Interest in being maintained on buprenorphine for OUD
* Plans to reside in current area for study period
* Achieving a study maintenance dose of >=8mg sublingual buprenorphine/naloxone
* Willing to comply with study protocol
* Have no clinically significant chronic medical or surgical disorders or conditions that are judged by the investigators to prevent participation

Exclusion Criteria:

* Medically contraindicated for buprenorphine, extended-release (XR)-buprenorphine (Sublocade), or suvorexant (as per medication labels)
* Pregnant or breast feeding
* Severe Diagnostic and Statistical Manual (DSM)-5 alcohol or benzodiazepine use disorder or evidence of alcohol/benzodiazepine physical dependence
* Have a known allergy to the study medications
* Past 30-day prescribed use of suvorexant for the indication of insomnia
* Current benzodiazepine or other prescribed medication for the indication of insomnia
* Urine sample testing positive for benzodiazepine at screening and admission to residential treatment
* Current narcolepsy, restless leg syndrome or sleep paralysis
* High risk for current sleep apnea
* Current (past 30-day) suicidal behaviors
* Severe hepatic or renal impairment

  * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3x upper limit of normal (ULN)
  * Total bilirubin >2x ULN
  * Creatinine >1.5x ULN
* Past year clinically-significant psychiatric condition judged to interfere with study participation
* Lack of access to stable housing (necessary for electronic pill dispenser charging)
* Have circumstances that would interfere with study participation (e.g., impending jail)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time | 3 nights during the initial residential phase and 1 night at the end of outpatient treatment
  Duration of nightly total sleep time in minutes, as measured by electroencephalography (EEG) and supplemented by actigraphy/photoplethysmography (e.g., if EEG malfunctions).
Buprenorphine compliance as assessed by the number of study days complying with buprenorphine treatment | 25 days across residential and outpatient treatment
  Buprenorphine compliance will be assessed by the number of study days complying with buprenorphine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Huhn, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No